CLINICAL TRIAL: NCT01012687
Title: A Single Dose, Two-Period, Two-Treatment, Two-Sequence Crossover Bioequivalency Study of Perindopril Erbumine Tablets 8 mg Under Fasting Conditions
Brief Title: Bioequivalency Study of Perindopril Erbumine 8 mg Tablet Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PERI-T8-PVFS-1
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: perindopril erbumine — 8 mg tablet
  Other Names: Aceon

SUMMARY:
The objective of this study was to prove the bioequivalence of Perindopril Erbumine 8 mg tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to perindopril or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 20 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States